CLINICAL TRIAL: NCT00130390
Title: Multi-center, Randomized, Double-Blind, Placebo-Controlled Trial of Nitazoxanide Tablets in the Treatment of Mild to Moderate Active Crohn's Disease in Adults
Brief Title: Study of Nitazoxanide Tablets in the Treatment of Mild to Moderate Active Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: terminated due to slow recruitment
Sponsor: Romark Laboratories L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RM01-2018
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — nitazoxanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): One nitazoxanide 500 mg tablet twice daily for 28 days
  Interventions: Drug: Nitazoxanide
- 2 (Placebo Comparator): One placebo tablet twice daily for 28 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nitazoxanide — One nitazoxanide 500 mg tablet twice daily for 28 days
  Other Names: Alinia
  Arms: 1
Other: Placebo — One placebo tablet twice daily for 28 days
  Arms: 2

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of nitazoxanide compared to a placebo in reducing the signs and symptoms of mild to moderate active Crohn's disease in adults.

DETAILED DESCRIPTION:
There is a significant need for a safe and effective treatment of Crohn's disease. It is recognized that bacteria in the gut lumen may have a role in the etiology and/or symptoms of this disease. Antimicrobials have often been used in treating Crohn's disease although their effectiveness has not been well established. Pro-inflammatory cytokines are also believed to play an important role in this disease. Nitazoxanide, a thiazolide anti-infective, is active in vitro against a broad spectrum of anaerobic bacteria, and it inhibits secretion of pro-inflammatory cytokines including IL-2, -4, -5, -6, -8, -10 and TNF alpha. The drug is also highly concentrated in the gastrointestinal tract. With these characteristics, nitazoxanide offers a unique approach to treatment of Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Diagnosis of Crohn's disease with colonic or perianal involvement confirmed by endoscopic, histologic and/or radiologic data.
* CDAI score ≥200 and ≤400.

Exclusion Criteria:

* Subjects known to have stool positive for Clostridium difficile toxin A or B, bacterial enteric pathogens, rotavirus, Cryptosporidium species (spp.), and/or ova/parasites.
* Evidence of bowel obstruction.
* Females that are pregnant, breast-feeding or not using birth control and are sexually active.
* Serious systemic disorders incompatible with the study.
* History of hypersensitivity to nitazoxanide or any inactive ingredient in the formulation.
* Uncontrolled gastro-intestinal bleeding.
* Evidence of intestinal abscess, non-perianal fistula or stricture.
* Patients who have received antibiotics in the past 7 days.
* Patients receiving >20 mg of prednisone, or its equivalent.
* Patients receiving Anucort-HC or rectal steroids.
* Patients receiving immunosuppressive therapy that has not been stabilized.
* Patients who have received TNF-alpha inhibitor treatments such as infliximab or other biological agents within three months prior to start of treatment.
* Patients with Crohn's disease confined to the esophagus, stomach and small bowel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2005-08; Primary Completion 2007-12 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Change in Crohn's Disease Activity Index (CDAI) | Day 14

SECONDARY OUTCOMES:
Clinical response; remission; change in C-reactive protein; reduction in steroid use; fistula response; change in Perianal Disease Activity Index (PDAI); change in plasma cytokine levels | Days 14 and 28

CONTACTS AND LOCATIONS:
Overall Officials: Maria Carrion, MD, Study Director — Romark Laboratories L.C.
Locations (13):
- United States (13):
  - Romark Laboratories, L.C., Tampa, Florida
  - Florida medical Clinic, P.A., Zephyrhills, Florida
  - Atlanta Gastroenterology, Marietta, Georgia
  - Atlanta Gastroenterology, Woodstock, Georgia
  - Gasteroenterology Associates, Baton Rouge, Louisiana
  - Minnesota Gastroenterology, P.A., Clinical Research Division, Plymouth, Minnesota
  - Long Island Clinical Research Associates, LLP, Great Neck, New York
  - Greater Cincinnati Gastroenterology Associates, Cincinnati, Ohio
  - Digestive Research & Infusion Institute, Mayfield Heights, Ohio
  - Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma
  - Memphis Gastroenterology Group, Germantown, Tennessee
  - Gastrointestinal Associates, LLC, Kingsport, Tennessee
  - Nashville Medical Research, Nashville, Tennessee